CLINICAL TRIAL: NCT01583283
Title: A Phase 1/2, Open-Label, Multicenter Study of ACY-1215 (Ricolinostat) in Combination With Lenalidomide and Dexamethasone for the Treatment of Relapsed or Relapsed/Refractory Multiple Myeloma
Brief Title: Study of ACY-1215 in Combination With Lenalidomide, and Dexamethasone in Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-MM-101
Record Dates: First submitted 2012-04-11; First posted 2012-04-24 (Estimated); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Relapsed; Refractory; Histone deacetylase inhibitors; Lenalidomide; Revlimid; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — ricolinostat; Histone Deacetylase Inhibitors; Lenalidomide; Dexamethasone; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACY-1215, Lenalidomide and Dexamethasone (Experimental): Open label dosing cohorts will evaluate oral ACY-1215 (doses ranging from 40 - 480 mg days 1-5, 8-12, 15-19) in combination with oral Lenalidomide (doses ranging from 15 - 25 mg days 1-21) and oral Dexamethasone (40 mg once weekly).
  Interventions: Drug: ACY-1215; Drug: lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: ACY-1215 — Dose escalation up to 480 mg administered orally on Days 1-5, 8-12 and 15-19 of a 28 day dosing schedule.
  Other Names: Histone deacetylase inhibitor
Drug: lenalidomide — Dosed on Days 1-21 of a 28 day cycle.
  Other Names: Revlimid
Drug: Dexamethasone — Dosed on Days 1, 8, 15 and 22 of a 28 day treatment cycle.
  Other Names: steroid

SUMMARY:
The purpose of this study is to determine the best dose of ACY-1215 in combination with lenalidomide and dexamethasone in patients with relapsed or relapsed/refractory multiple myeloma. Once determined, the purpose of this study will be to determine the efficacy of ACY-1215 in combination with lenalidomide and dexamethasone in patients with relapsed multiple myeloma who have had 1-3 prior therapies and who are not lenalidomide-refractory.

DETAILED DESCRIPTION:
This is phase 1, single-arm, multicenter, open-label study in patients with relapsed or relapsed/refractory MM. The study employs a sequential group dose-escalation design to determine the DLT and MTD of ACY-1215 in combination with lenalidomide and dexamethasone, all administered orally (PO). The safety, tolerability, single- and multiple-dose PK, pharmacodynamics, and anti-tumor activity of ACY 1215 in combination with lenalidomide and dexamethasone also will be evaluated.

Each cohort will enroll 3 patients. Study drug doses will be escalated sequentially after the Safety Review Committee (SRC) reviews safety data collected in C1 (28 days) from patients enrolled at the current dose level as well as emerging data from ongoing studies of ACY-1215. If there are no DLTs (as defined in Section 5.2.6) during C1 or concerns based on data from other ongoing studies, the study will proceed with dose escalation to the next cohort following safety data review by the SRC. If 1 of 3 patients has a DLT, then up to 3 additional patients will be enrolled in that cohort; if none of the additional 3 patients experience a DLT during C1, escalation may then continue to the next cohort following SRC review. If 2 or more patients have DLTs during C1, the DLT dose level will have been reached.

The MTD is defined as the dose level immediately below the DLT dose level. A total of up to 6 additional patients may be enrolled at the MTD or other appropriate dose level to obtain additional AE, PK, pharmacodynamic, and anti-tumor activity data on ACY 1215 in combination with lenalidomide and dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or Relapsed/Refractory MM with progressive disease (PD) according to IMWG.
* Received at least 1 prior line of therapy for MM (Phase 1)
* Secretory MM for which the patient previously received 1-3 prior lines of therapy (Phase 2).
* Able to provide written consent
* Not a candidate for autologous stem cell transplant (ASCT) or declined option.
* ≥18 years of age
* Karnofsky Performance Status score ≥ 70
* Adequate bone marrow reserve as evidenced by ANC > 1.0x10^9/L;Platelet > 50x10^9/L
* Creatinine Clearance of ≥ 50 mL/min
* Adequate hepatic function as evidenced by serum bilirubin values < 2.0 mg/dL; ALT and/or AST < 3xULN.
* Corrected serum calcium ≤ ULN
* Recovered from the effects of any prior systemic therapy or radiotherapy for Multiple Myeloma
* Able to take acetylsalicylic acid (ASA) (81 or 325 mg) daily as prophylactic anticoagulation. Patients intolerant to ASA may use low molecular weight heparin. Lovenox is recommended. Coumadin will be allowed provided the patient is fully anticoagulated, with an INR of 2 or 3.
* Agreement to participate in RevAssist® Program
* Female of childbearing potential must have a negative serum or urinary pregnancy test with a sensitivity of at least 50 mIU/mL 10-14 days prior to and again within 24 hours of prescribing lenalidomide for Cycle 1 and must either commit to continued abstinence or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method at the same time, at least 28 days prior to taking lenalidomide. Also agree to ongoing pregnancy testing.
* If male, including those who have had a vasectomy, must agree to use a latex condom during any sexual contact with a female of childbearing potential.

Exclusion Criteria:

* Received any of the following antitumor therapies

  * Radiotherapy or systemic therapy within 2 weeks of Cycle 1 Day 1 (C1D1)
  * Investigational or biologic therapies within 3 weeks of C1D1
  * Prior peripheral ASCT within 12 weeks of C1D1
  * Prior allogeneic stem cell transplant
  * Prior treatment with a histone deacetylase (HDAC) inhibitor
* Presence of an active systemic infection requiring treatment.
* History of other malignancies unless a.) the patient has undergone definitive treatment more than 5 years prior and is without evidence of recurrent malignant disease or b.) had basal or squamous cell carcinoma of the skin; superficial carcinoma of the bladder; carcinoma of the prostate with current prostat specific antigen < 0.1 ng/mL; ductal carcinoma in situ; or cervical intraepithelial neoplasia.
* Known or suspected human immunodeficiency virus (HIV), hepatitis B surface antigen-positive status or known or suspected active hepatitis C infection.
* If female, is lactating.
* History of significant cardiovascular, neurological, endocrine, gastrointestinal, respiratory, or inflammatory illness that could preclude study participation, pose an undue medical hazard, or interfere with the interpretation of the study results, including but not limited to congestive heart failure (NYHA Class 3 or 4), unstable angina; cardiac arrhythmia, recent (within past 6 months) myocardial infarction or stroke; uncontrolled hypertension; diabetes mellitus with >2 episodes of ketoacidosis in the preceding 12 months, COPD requiring >2 hospitalizations in preceding 12 months
* QTcF > 480 msec, family or personal history of long QTc syndrome or ventricular bigeminy; previous history of drug-induced QTc prolongation or the need for medications known or suspected of producing prolonged QTc intervals on ECG
* Current enrollment in another clinical trial involving treatment and/or is receiving an investigational agent for any reason
* Documented plasma cell leukemia or known amyloidosis. (Plasma cell leukemia is defined as the presence of >20% plasma cells in the peripheral blood and an absolute plasma cell count of ≥2000 muL
* Known hypersensitivity to thalidomide or lenalidomide.
* History of erythema nodosum characterized by desquamating rash while taking thalidomide or similar drugs.
* Non-secretory or oligo-secretory Multiple Myeloma (Phase II only; such disease is permissible in Phase I).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-07-12 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-24 (Actual)

PRIMARY OUTCOMES:
To determine DLT of ACY-1215 administered in combination with lenalidomide and dexamethasone in patient with relapsed/refractory MM | up to 7 years
  Number of participants with Dose Limiting Toxicity (DLT)
To determine MTD of ACY-1215 administered in combination with lenalidomide and dexamethasone in patient with relapsed/refractory MM | up to 7 years
  Maximum Tolerated Dose is defined as the dose level immediately below the DLT dose level.
Objective Response Rate of ACY-1215 | up to 7 years
  The objective response rate is the proportion of subjects achieving an investigator conformed partial response (PR) or better, to treatment according to IMWG (International Myeloma Working Group).

SECONDARY OUTCOMES:
Duration of Response | Up to approximately 7 years
  The duration of response is defined as the time (in weeks) from the date of the first documentation of objective response to the first documentation of objective tumor progression or death on study due to any cause, whichever comes first.
Adverse Events (AEs) | From enrollment until at least 28 days after completion of study treatment
  Number of participants with adverse event
Disease Control Rate | Up to approximately 7 years
  Disease control rate is defined as the proportion of subjects with a response (Unconfirmed or Confirmed) of SD or better, more specifically sCR, CR, VGPR, PR, MR, or SD respectively.
Progression-free Survival | Up to approximately 7 years
  PFS is defined as the time (in weeks) from the date of first dose to the date of first documentation of disease progression or death on study due to any cause, whichever comes first.
Evaluate the pharmacodynamics of ACY-1215 in combination with lenalidomide and dexamethasone in patients with relapsed or relapsed/refractory MM | up to 28 days
  Exposure-response of ACY-1215 in combination with lenalidomide and dexamethasone, including biomarkers relating to intracellular protein acetylation, levels of proteins, messenger ribonucleic acid (mRNA) and microRNA expression profiles will be analyzed for potential relationships.
Pharmacokinetic- Cmax | up to 28 days
  Maximum serum concentration
Pharmacokinetic- Cmin | up to 28 days
  Minimum observed concentration
Pharmacokinetic- Tmax | up to 28 days
  Time to maximum serum concentration
Pharmacokinetic- AUC | up to 28 days
  Area under the plasma concentration time curve
Pharmacokinetic- t1/2 | up to 28 days
  Serum half-life

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- United States (5):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of North Carolina, Chapel Hill, North Carolina
  - Sarah Cannon Research Institute Drug Development Unit, Nashville, Tennessee
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Clinical Study Report

REFERENCES:
- [Background] Tamang D, et al. Tubulin Hyper-Acetylation In Blood Lymphocytes: Pharmacodynamic (PD) Biomarker For The Selective Histone Deacetylase (HDAC) 6 Inhibitor ACY-1215 In Multiple Myeloma (MM) Patients. Presented at American Society of Hematology 2013, December 7-10, 2013, New Orleans, LA. Abstract No. 3219.
- [Result] Yee AJ, Bensinger WI, Supko JG, Voorhees PM, Berdeja JG, Richardson PG, Libby EN, Wallace EE, Birrer NE, Burke JN, Tamang DL, Yang M, Jones SS, Wheeler CA, Markelewicz RJ, Raje NS. Ricolinostat plus lenalidomide, and dexamethasone in relapsed or refractory multiple myeloma: a multicentre phase 1b trial. Lancet Oncol. 2016 Nov;17(11):1569-1578. doi: 10.1016/S1470-2045(16)30375-8. Epub 2016 Sep 17. PMID 27646843
- [Result] Yee, Andrew & Bensinger, William & Voorhees, Peter & Berdeja, Jesus & Richardson, Paul & Supko, Jeffrey & Tamang, David & Jones, Simon & Wheeler, Catherine & Markelewicz, Robert & Raje, Noopur. (2015). Ricolinostat (ACY-1215), the First Selective HDAC6 Inhibitor, in Combonation with Lenalidomide and Dexamethasone in Patients with Relapsed and Relapsed-and-Refractory Multiple Myeloma: Phase 1b Results (ACE-MM-101 Study). Blood 2015; 126(23): 3055-3055.doi: 10.1182/blood.v126.23.3055.3055.
- [Result] Yee, Andrew & Voorhees, Peter & Bensinger, William & Berdeja, Jesus & Supko, Jeffrey & Richardson, Paul & Tamang, David & Jones, Simon & Patrick, Gretchen & Wheeler, Catherine & Raje, Noopur. (2014). Ricolinostat (ACY-1215), a Selective HDAC6 Inhibitor, in Combination with Lenalidomide and Dexamethasone: Results of a Phase 1b Trial in Relapsed and Relapsed Refractory Multiple Myeloma. Blood 2014; 124 (21): 4772-4772. doi:10.1182/blood.v124.21.4772.4772.
- [Result] RICOLINOSTAT (ACY-1215), THE FIRST SELECTIVE HISTONE DEACETYLASE 6 INHIBITOR, IS ACTIVE AND WELL TOLDERATED IN COMBINATION WITH LENALIDOMIDE OR BORTEZOMIB IN PATIENTS WITH REFRACTORY MYELOMA Raje N. EHA ePoster Jun 13, 2014; 53804 P358 https://library.ehaweb.org/eha/2014/19th/53804/noopur.raje.ricolinostat.28acy-121529